CLINICAL TRIAL: NCT05159453
Title: A Randomised, Multiple-Dose, Single Period, Phase II/III Dose Response Study to Examine Transdermal Human Insulin in Adult Diabetic Patients
Brief Title: Dose Response Study of Transdermal Human Insulin in Patients
Acronym: LEVPS
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Transdermal Delivery Solutions Corp (Industry)
Collaborators: Langford Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEV201-D-120121
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Glucose, High Blood
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Intervention Model Description: Single group, crossover study of insulin supplementation beginning with 2 weeks monitoring of response to injected dosing, crossover to transdermal dosing, then back to injected dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Main Experimental (Experimental): Type 2 Diabetic patients regulating blood glucose with daily injections as basal and/or post-prandial interventions. Patients will receive transdermal product formulated at 100 IU/mL of equivalent International Units of Human Insulin dosed at the same amount as current injected therapies with timing adjusted for the Absorption, Distribution, Metabolism & Elimination (ADME) of human insulin with maximum effect at 3 hours post dose so mid morning before lunch, late afternoon before dinner and before bedtime.
  Interventions: Biological: Human Insulin; Device: Finger-actuated, Metered Pump Sprayer

INTERVENTIONS:
Biological: Human Insulin — International Unit for International Unit exchange of transdermally delivered Human Insulin for injected Human Insulin or combinations of basal and fast-acting insulins.
  Other Names: Humulin(R); Novolin(R)
Device: Finger-actuated, Metered Pump Sprayer — Stock, pharmaceutical grade High Density Polyethylene (HDPE) bottle and HDPE nylon and stainless steel finger-actuated pump sprayer delivering 0.2 mL per pump.

SUMMARY:
A 21-Day open label study of transdermally delivered human insulin in Type 2 Diabetics as measured by response of down modulation of glucose after dosing of Insulin as compared to historic patient response to injected insulins.

DETAILED DESCRIPTION:
A 21-Day open label study of transdermally delivered human insulin in 30 Type 2 Diabetics is anticipated. Well-managed Type 2 Diabetics will be added to the protocol from the patient census of practicing diabetologists and family practitioners, with preference given to patients already using a wearable Continuous Glucose Monitor (CGM) system. Once added to the protocol, Subjects will be monitored via CGM for two weeks before change of dose form. Subjects will be required to calibrate the CGM against finger-stick blood sampling and to poll the monitor sensor at least every 8 hours during the 42 days of monitoring including the 21-days on-transdermal-dose study period to ensure continuity of interstitial glucose measurement. Subjects will be monitored for 7 days after the last transdermal dose to monitor interchangeability of the dose forms.

Once baseline data is collected, Subjects will exchange transdermal dosing on a Unit for Unit basis. Trial materials will be formulated to a concentration of 100 IUs per mL and dispensed via 0.2 mL metered, finger-actuated pump sprayer, with each pump delivering 20 IUs of Human Insulin to the skin. If a patient, for example is currently using 120 IUs per day, 40 IUs basal insulin and 80 IUs Insulin Aspart, 120 IUs or 6 sprays would be used.

The study nurse will contact each subject every day of the study to answer questions and encourage compliance with the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Type 2 Diabetes Mellitus ("T2D") Patients on Insulin Replacement therapy not administered via implanted pump well-managing p.r.n as defined by serum glucose ranging between 85 and 200 mg/dL and no more than 1 hypoglycemic or serious hypoglycemic event within the last 9 months.
2. 25 and 75 years of age, inclusive.
3. The subject is willing and able to read and understand the Subject Information Sheet and provide written informed consent.
4. The subject has a body mass index (BMI) within 18-50 kg/m2.
5. The subject is in otherwise good health as determined by medical history and physical examination.
6. The subject's normal insulin dose ranges from between 10 to 200 IU per dose.
7. The subject must agree to continue with daily serum glucose testing by means of a wearable blood glucose monitor for the pharmacodynamic assessments that the investigators have continuous access to via daily downloads.
8. The subject is willing and able to comply with all testing and requirements defined in the protocol.
9. The subject is willing and able to return to the study site for all visits.

Exclusion Criteria:

1. The subject has any relevant deviations from normal other than blood glucose in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator.
2. The subject has had more than 2 hypoglycemic events in the last month.
3. The subject's normal insulin dose is less than 10 and more than 200 IUs.
4. Subjects receiving Insulin from an implanted or external insulin pump system.
5. The subject has had a clinically significant illness or surgical procedure within 30 days preceding entry into this study.
6. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease other than T2D.
7. The subject has a known allergy or history of hypersensitivity to Human Insulin or similar modified Insulin compounds.
8. The subject has used any prescription medication that may interfere with the evaluation of study medication.
9. The subject has donated or lost a significant volume of blood (>450 mL) within four (4) weeks of the study, and subject's Hemoglobin concentration and hematocrit have not returned to within 5% of normal.
10. The subject has a history of substance abuse or a current positive urine drug screen or urine alcohol test.
11. Alcohol consumption greater than community norms (i.e. more than 21 standard drinks per week for males).
12. Subjects who have received an investigational drug or have used an investigational device in the 30 days prior to study entry.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Glucose Time in Range for Study Participants | 21 Days
  Number of Participants who manage blood glucose in study participants to between 70 and 200 mg Glucose / dL.

SECONDARY OUTCOMES:
Avoidance of Hypoglycemia in Study Participants | 21 days.
  Number of study participants that manage blood glucose in study participants to more than 50 mg/dL for 86% of the 21-days-on-dose of the study period
Skin Safety in Study Participants | 21 days dosing plus 7 days post dose follow-up.
  Measure of skin irritation above level 1 - erythema & edema - according to the The Organisation for Economic Co-operation and Development (OECD) Guideline for Testing of Chemicals No. 404, adopted 17th July, 1992: "Acute Dermal Irritation/Corrosion"

CONTACTS AND LOCATIONS:
Overall Officials: William D. Kirsh, D.O., Principal Investigator — University of Miami
Locations (1):
- Langford Research Institute, Palm Beach Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: No